CLINICAL TRIAL: NCT03663764
Title: Hypofractionated Radiotherapy Combined With Concurrent Weekly Chemotherapy and Thymosin α1 in Patients With Unresectable or Recurrent Thymic Epithelial Tumor: A Prospective, Single-arm Phase II Study
Brief Title: Hypofractionated Chemoradiotherapy and Thymosin α1 in Unresectable or Recurrent Thymic Epithelial Tumor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-1042
Record Dates: First submitted 2018-09-04; First posted 2018-09-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Thymoma and Thymic Carcinoma
Keywords: Unresectable or Recurrent Thymoma and Thymic Carcinoma; Hypofractionated Chemoradiotherapy; Thymosin a1
MeSH Terms: conditions — Thymoma | interventions — Radiation Dose Hypofractionation; Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Expeiment (Experimental): HRT using the IMRT technique was administered. For patients with limited pulmonary or pleural metastases (≤3 lesions), stereotactic body radiation therapy (SBRT) could be used.
  All patients received weekly docetaxel(25mg/㎡) and nedaplatin or cisplatin (25mg/㎡), each of 1 day's duration, concurrently with hypofractionated radiotherapy .
  Meanwhile they received weekly thymosin a1(1.6mg) during and within 2 months after the end of chemoradiotherapy.
  Interventions: Drug: Thymosin a1; Radiation: hypofractionated radiotherapy; Drug: concurrent chemoradiotherapy

INTERVENTIONS:
Drug: Thymosin a1 — All patients received weekly thymosin a1(1.6mg) during and within 2 months after the end of chemoradiotherapy.
Radiation: hypofractionated radiotherapy — HRT using the IMRT technique was administered. For patients with limited pulmonary or pleural metastases (≤3 lesions), stereotactic body radiation therapy (SBRT) could be used.
Drug: concurrent chemoradiotherapy — All patients received weekly docetaxel(25mg/㎡) and nedaplatin or cisplatin (25mg/㎡), each of 1 day's duration, concurrently with hypofractionated radiotherapy .

SUMMARY:
This phase II study was to assess the efficacy and toxicity of hypofractionated radiotherapy (HRT) combined with weekly docetaxel/platinum and thymosin α1 in patients with unresectable or recurrent thymic epithelia tumors (TETs).

DETAILED DESCRIPTION:
HRT using the IMRT technique was administered. For patients with limited pulmonary or pleural metastases (≤3 lesions), stereotactic body radiation therapy (SBRT) could be used.

All patients received weekly docetaxel(25mg/㎡) and nedaplatin or cisplatin (25mg/㎡), each of 1 day's duration, concurrently with hypofractionated radiotherapy .

Meanwhile they received weekly thymosin a1(1.6mg) during and within 2 months after the end of chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of thymoma, thymic carcinoma or thymic endocrine tumors.
* Patients have measurable or evaluable lesions based on the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Unresectable disease or recurrent intrathoracic disease which could be encompassed within radiation fields.
* White blood cell count ≥4×109 /L, neutrophile granulocyte count≥1.5×109 /L, platelet count≥100×109 /L, hemoglobin ≥100 g /L, serum creatinine and bilirubin 1.5 times less than the upper limits of normal (ULN),aminotransferase two times less than the ULN.
* FEV1 >0.8 L
* CB6 within normal limits
* Patients and their family signed the informed consents

Exclusion Criteria:

* Previous or recent another malignancy, except for nonmelanoma skin cancer or cervical cancer in situ.
* Any contraindication for chemotherapy or radiotherapy(such as a myocardial infarction within 6 months,immunosuppressive therapy,symptomatic heart disease,including unstable angina pectoris, congestive heart failure,and uncontrolled arrhythmia).
* Malignant pleural effusion or pericardial effusion.
* Weight loss >10% within the past 3 months.
* Recruited in other clinical trials within 30 days
* Drug addiction, long-term alcohol abuse and AIDS patients.
* Uncontrollable epileptic attack or psychotic patients without self-control ability.
* Severe allergy or idiosyncrasy.
* Not suitable for this study judged by researchers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2018-08-13 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | 2 years

SECONDARY OUTCOMES:
Quality of Life score | 1 year
  EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer) core questionnaire
Overall Survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Professor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Detterbeck F, Youssef S, Ruffini E, Okumura M. A review of prognostic factors in thymic malignancies. J Thorac Oncol. 2011 Jul;6(7 Suppl 3):S1698-704. doi: 10.1097/JTO.0b013e31821e7b12. No abstract available. PMID 21847050
- [Background] Detterbeck FC, Nicholson AG, Kondo K, Van Schil P, Moran C. The Masaoka-Koga stage classification for thymic malignancies: clarification and definition of terms. J Thorac Oncol. 2011 Jul;6(7 Suppl 3):S1710-6. doi: 10.1097/JTO.0b013e31821e8cff. No abstract available. PMID 21847052
- [Background] Gao L, Wang C, Fang W, Zhang J, Lv C, Fu S. Outcome of multimodality treatment for 188 cases of type B3 thymoma. J Thorac Oncol. 2013 Oct;8(10):1329-34. doi: 10.1097/JTO.0b013e31829ceb50. PMID 24457243
- [Background] Marx A, Strobel P, Badve SS, Chalabreysse L, Chan JK, Chen G, de Leval L, Detterbeck F, Girard N, Huang J, Kurrer MO, Lauriola L, Marino M, Matsuno Y, Molina TJ, Mukai K, Nicholson AG, Nonaka D, Rieker R, Rosai J, Ruffini E, Travis WD. ITMIG consensus statement on the use of the WHO histological classification of thymoma and thymic carcinoma: refined definitions, histological criteria, and reporting. J Thorac Oncol. 2014 May;9(5):596-611. doi: 10.1097/JTO.0000000000000154. PMID 24722150
- [Background] Guerrera F, Rendina EA, Venuta F, Margaritora S, Ciccone AM, Novellis P, Novero D, Anile M, Bora G, Rena O, Casadio C, Mussi A, Evangelista A, Ruffini E, Lucchi M, Filosso PL. Does the World Health Organization histological classification predict outcomes after thymomectomy? Results of a multicentre study on 750 patients. Eur J Cardiothorac Surg. 2015 Jul;48(1):48-54. doi: 10.1093/ejcts/ezu368. Epub 2014 Sep 21. PMID 25246487
- [Background] Onuki T, Ishikawa S, Yamamoto T, Ito H, Sakai M, Onizuka M, Sakakibara Y, Iijima T, Noguchi M, Ohara K. Pathologic radioresponse of preoperatively irradiated invasive thymomas. J Thorac Oncol. 2008 Mar;3(3):270-6. doi: 10.1097/JTO.0b013e3181653c8c. PMID 18317070
- [Background] Bretti S, Berruti A, Loddo C, Sperone P, Casadio C, Tessa M, Ardissone F, Gorzegno G, Sacco M, Manzin E, Borasio P, Sannazzari GL, Maggi G, Dogliotti L; Piemonte Oncology Network. Multimodal management of stages III-IVa malignant thymoma. Lung Cancer. 2004 Apr;44(1):69-77. doi: 10.1016/j.lungcan.2003.09.022. PMID 15013585
- [Background] Wright CD, Choi NC, Wain JC, Mathisen DJ, Lynch TJ, Fidias P. Induction chemoradiotherapy followed by resection for locally advanced Masaoka stage III and IVA thymic tumors. Ann Thorac Surg. 2008 Feb;85(2):385-9. doi: 10.1016/j.athoracsur.2007.08.051. PMID 18222230
- [Background] Korst RJ, Bezjak A, Blackmon S, Choi N, Fidias P, Liu G, Marx A, Wright C, Mock S, Rutledge JR, Keshavjee S. Neoadjuvant chemoradiotherapy for locally advanced thymic tumors: a phase II, multi-institutional clinical trial. J Thorac Cardiovasc Surg. 2014 Jan;147(1):36-44, 46.e1. doi: 10.1016/j.jtcvs.2013.08.061. Epub 2013 Oct 15. PMID 24139613
- [Background] Venuta F, Rendina EA, Pescarmona EO, De Giacomo T, Vegna ML, Fazi P, Flaishman I, Guarino E, Ricci C. Multimodality treatment of thymoma: a prospective study. Ann Thorac Surg. 1997 Dec;64(6):1585-91; discussion 1591-2. doi: 10.1016/s0003-4975(97)00629-2. PMID 9436540
- [Background] Lucchi M, Mussi A, Basolo F, Ambrogi MC, Fontanini G, Angeletti CA. The multimodality treatment of thymic carcinoma. Eur J Cardiothorac Surg. 2001 May;19(5):566-9. doi: 10.1016/s1010-7940(01)00666-2. PMID 11343932
- [Background] Rea F, Sartori F, Loy M, Calabro F, Fornasiero A, Daniele O, Altavilla G. Chemotherapy and operation for invasive thymoma. J Thorac Cardiovasc Surg. 1993 Sep;106(3):543-9. PMID 8361199
- [Background] Yokoi K, Matsuguma H, Nakahara R, Kondo T, Kamiyama Y, Mori K, Miyazawa N. Multidisciplinary treatment for advanced invasive thymoma with cisplatin, doxorubicin, and methylprednisolone. J Thorac Oncol. 2007 Jan;2(1):73-8. doi: 10.1097/JTO.0b013e31802bafc8. PMID 17410014
- [Background] Goldstein AL. History of the discovery of the thymosins. Ann N Y Acad Sci. 2007 Sep;1112:1-13. doi: 10.1196/annals.1415.045. Epub 2007 Jun 28. PMID 17600284
- [Background] Garaci E, Pica F, Sinibaldi-Vallebona P, Pierimarchi P, Mastino A, Matteucci C, Rasi G. Thymosin alpha(1) in combination with cytokines and chemotherapy for the treatment of cancer. Int Immunopharmacol. 2003 Aug;3(8):1145-50. doi: 10.1016/S1567-5769(03)00053-5. PMID 12860169
- [Background] Jiang J, Wang X, Tian J, Li L, Lin Q. Thymosin plus cisplatin with vinorelbine or gemcitabine for non-small cell lung cancer: A systematic review and meta-analysis of randomized controlled trials. Thorac Cancer. 2011 Nov;2(4):213-220. doi: 10.1111/j.1759-7714.2011.00057.x. PMID 27755854